CLINICAL TRIAL: NCT05907733
Title: Brain-derived Neurotrophic Factor (BDNF) Single Nucleotide Gene Polymorphism and Nerve Growth Factor as Risk Factors That Increase Severity of Allergic Rhinitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud Kadry, lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-04-09PD
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Genotyping. — 5 ml biood withdrawen by venipuncture in EDTA tube DNA extraction will be done after centrifucation and used for quantatitive Real-time polymerase chain reaction.
  Other Names: Measurement of Nerve growth factor serum level

SUMMARY:
Allergic diseases such as asthma, allergic rhinitis (AR) and atopic dermatitis affect more than 25% of the world population and are the leading cause of illness in children. The complex interplay between genetic, environmental and immunological risk factors results in the manifestation of allergic diseases . The pathological presentation of allergic disease involves the activation of both the innate and adaptive immune systems, resulting in a multifaceted response in specific target tissues such as the airways . This response results in the recruitment of inflammatory cells to target tissues and the production of specific IgE antibodies, cytokines and other inflammatory mediators [11], [12]. It is well established that allergic inflammation triggers neuronal dysfunction, which activates specific inflammatory mechanisms, potentially leading to structural changes in the diseased tissue . Neurotrophins are a family of structurally related proteins initially discovered to be involved in regulating neuronal development and now known to govern both peripheral and central nerve growth.

BDNF is a secretory protein belonging to the neurotrophin family and is involved in a range of neural processes during human development [19], [20]. In the early stages of development BDNF is essential for neurogenesis, survival and maturation of neuronal pathways. In the adult, alongside neurotransmitters, hormones and other neurotrophins, BDNF maintains synaptic plasticity, dendritic growth and the consolidation of long-term memory. The biological effect of BDNF is mediated via its binding to the trkB receptor. The activation of these receptors on eosinophils may be important in regulating the inflammatory cascade leading to allergic disease [15], [24]. Neurotrophin mediated activation of bronchial eosinophils might therefore play a role in the regulation of eosinophilic inflammation in allergic asthma .

The BDNF gene is located on chromosome 11p13 and is alternatively spliced resulting in several different transcripts [26]. Genetic polymorphisms in BDNF have been associated with allergic phenotypes such atopic dermatitis [27] and asthma [28], [29], [30], [31] in different populations. The functional polymorphism rs6265 (Val66Met) has been shown to regulate intracellular trafficking and affect the secretion of BDNF [32]. Nerve growth factor (NGF), a neurotrophin that is expressed in the glandular, nasal epithelium, and peripheral nerves in the nasal mucosa, has been shown to induce biochemical and structural changes in nerves that can lead to hyper-responsiveness [33], [34], [35] The biological effects of neurotrophins are mediated by binding either to the high-affinity tyrosine kinase (trk) receptors or to the low-affinity receptors known as pan-neurotrophin receptor p-75.

ELIGIBILITY:
Inclusion Criteria:

* The chronic AR patients on anti-allergic .

Exclusion Criteria:

* The chronic AR patients on anti-allergic therapy will be excluded.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on 50 patients 30 patients diagnosed as a clinical disease of AR according to the diagnostic criteria of AR based on, its Impact on Asthma criteria, the patient's history of allergic symptoms, and allergy test results using the ImmunoCAP system.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
BDNF gene single nucleotide polymorphism with Allergic rhinitis risk | 2 months
  will measure in blood
Nerve growth factor serum level | 2 months
  will measure in blood for the risk of Allergic rhinitis.
IL-1 serum level | 2 months
  will measure in blood for the risk of Allergic rhinitis.
C-reactive protein serum level | 2 months
  will measure in blood for the risk of Allergic rhinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nathan RA. The burden of allergic rhinitis. Allergy Asthma Proc. 2007 Jan-Feb;28(1):3-9. doi: 10.2500/aap.2007.28.2934. PMID 17390749
- [Background] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D; World Health Organization; GA(2)LEN; AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008 Apr;63 Suppl 86:8-160. doi: 10.1111/j.1398-9995.2007.01620.x. No abstract available. PMID 18331513
- [Background] Devereux G. The increase in the prevalence of asthma and allergy: food for thought. Nat Rev Immunol. 2006 Nov;6(11):869-74. doi: 10.1038/nri1958. PMID 17063187
- [Background] Vercelli D. Discovering susceptibility genes for asthma and allergy. Nat Rev Immunol. 2008 Mar;8(3):169-82. doi: 10.1038/nri2257. PMID 18301422